CLINICAL TRIAL: NCT06856746
Title: Smartphone-based Utility of the Vestibulo-ocular Reflex: a Pilot Clinical Study
Brief Title: Smartphone-based Utility of the Vestibulo-ocular Reflex
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Principal Investigator, Bradley Kesser, MD, Department Vice-Chair, University of Virginia
Other Study IDs: HSR230265; 1R41DC022209-01 (NIH)
Record Dates: First submitted 2025-02-12; First posted 2025-03-04 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-04

CONDITIONS: Vestibulo-Ocular Reflex (VOR) Dysfunction; Vestibular Function Tests; Vestibular Function Disorder; mHealth Application
Keywords: Vestibular Dysfunction; Gaze Stabilization Test (GST); Vestibulo-Ocular Reflex (VOR); mHealth Vestibular Testing
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Unilateral vestibular dysfunction (UVD): This group includes with unilateral peripheral vestibular dysfunction identified via the Electronic Medical Record (EMR) and meet the following study criteria:
  Inclusion criteria:
  * > 18 y/o
  * Willingness and ability to comply with scheduled visits and study procedures.
  * History of unilateral vestibular dysfunction (>49% asymmetry on bithermal binaural caloric testing) OR surgical ablation of vestibular end organ or nerve, such as via resection of unilateral vestibular schwannoma or labyrinthectomy)
  Exclusion criteria:
  * No history of vestibular dysfunction
  * History of underlying cervical musculoskeletal disease that restricts the neck
  * History of cervical dysfunction that prevented them from moving their head, severe visual impairment or blind spots in the field, or central nervous system disorder
- Healthy volunteers: This group includes with those without a history of unilateral peripheral dysfunction (UVD) and meet the following study criteria:
  Inclusion criteria:
  * 18 y/o
  * Willingness and ability to comply with scheduled visits and study procedures
  Exclusion criteria:
  * History of vestibular dysfunction
  * History of uncorrected vision
  * History of underlying cervical musculoskeletal disease that restricts the neck
  * History of cervical dysfunction that prevented them from moving their head, severe visual impairment or blind spots in the field, or central nervous system disorder

SUMMARY:
The goal of this observational study is to evaluate whether a novel smartphone-based (mHealth) application can accurately assess gaze stability and vestibulo-ocular reflex (VOR) function in adults with vestibular dysfunction. This pilot clinical ststudy includes adult participants with and without unilateral peripheral vestibular dysfunction to determine the feasibility of a mobile-based assessment of gaze stabilization.

The main questions it aims to answer are:

1. Can a prototype mHealth application accurately measure outcomes associated with standard dynamic gaze stabilization tests (e.g., static visual acuity, perception time, and maximal head velocity measurements)?
2. How well does a prototype mHealth application identify patients with unilateral peripheral vestibular dysfunction when compared to healthy volunteers?
3. Does a prototype mHealth application differ in identifying patients with unilateral peripheral vestibular dysfunction when compared to a commercially-available computer system that uses a gold-standard head-mounted sensor for gaze stabilization testing (GST)?

Participants will:

Perform the well-established GST protocol using a commercially-available computer system that uses a gold-standard head-mounted sensor Perform the well-established GST protocol a novel mHealth application

The following outcomes will be measured:

1. Standard visual acuity (SVA): The smallest readable target based on the user's best-aided vision
2. A perception time test (PTT): The shortest time a target can be accurately identified
3. A dynamic gaze stability test (GST): The maximal head velocity at which a patient can accurately identify the orientation of a presented visual target

This pilot clinical study will provide evidence to further support the use of mobile technology as a low-cost, accessible alternative for vestibular function assessment, particularly for patients in resource-limited settings.

DETAILED DESCRIPTION:
Background & Rationale Vestibular dysfunction is a common condition affecting over a third of U.S. adults over the age of 40. It significantly increases the risk of falls, especially in those experiencing dizziness, where the odds of falling are increased 12-fold. Current best practices recommend vestibular rehabilitation, which includes gaze stability exercises designed to improve balance and reduce fall risk. However, many individuals, particularly those relying on home-based therapy or telehealth, face challenges in accessing objective assessments of their vestibulo-ocular reflex (VOR) contribution to gaze stabilization.

As telehealth has expanded rapidly in response to the COVID-19 pandemic, there is an increasing need for remote, real-time VOR teleassessments that can provide clinicians and patients with quantifiable, velocity-specific gaze stability data. While some computer-based remote VOR assessment tools exist, they often suffer from limitations in user satisfaction and accuracy. The Gaze Stabilization Test (GST), developed by Goebel et al., provides clinicians with velocity-specific data associated with the VOR's contribution to gaze stabilization. However, this test is typically performed in a clinical setting with specialized equipment, limiting access for many patients.

This pilot clinical study aims to validate a mHealth application (mVOR) prototype as a low-cost, accessible alternative to traditional VOR assessments. By leveraging the head- and eye-tracking capabilities of modern smartphones, this proof-of-concept prototype seeks to provide a novel, mobile-based framework for measuring visual acuity, head velocity, and gaze estimation in patients undergoing vestibular rehabilitation.

Study Objectives & Hypothesis

Primary Objectives:

To determine whether a prototype mHealth application can accurately assess static visual acuity, perception time, and maximal head velocity in individuals with unilateral peripheral vestibular dysfunction (UVD).

To compare the accuracy of the mVOR application against a commercially-available, in-office GST system that identifies patients with UVD.

Hypothesis:

The investigators hypothesize that by using the native head and eye-tracking capabilities of smartphones, one can obtain gaze stability (GST) measurements using a mobile platform that provides visual acuity and velocity-specific data comparable to a commercially-available, in-office GST system.

If validated, the mVOR could serve as an platform for effective, low-cost alternatives for telemonitoring vestibular function and enhancing remote rehabilitation programs for individuals with balance disorders.

Anticipated sample size: 50 (25 healthy volunteers and 25 patients with UVD)

Data Analysis

Within-group comparisons:

Paired t-tests or Wilcoxon Signed-Rank tests (depending on data distribution) will compare participants' GST and mVOR scores.

Between-group comparisons:

Independent t-tests or Mann-Whitney U tests will compare UVD vs. healthy volunteer group.

ROC Curve Analysis:

Receiver Operating Characteristic (ROC) curves will assess the accuracy of mVOR vs. computerized GST in distinguishing patients with UVD

Potential Benefits & Clinical Significance Increased Accessibility: The mVOR app provides an affordable, mobile alternative to in-office based GST system, expanding access to vestibular rehabilitation.

Telehealth & Home Monitoring: This study could support remote vestibular assessments, particularly for patients in rural or underserved communities.

Clinical Validation: If the mVOR performs comparably to the in-office based GST, it may be integrated into clinical practice as a validated tool for assessing vestibular function.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Able to provide informed consent
* Normal or corrected-to-normal vision (e.g., with glasses or contact lenses)
* Able to sit upright and follow instructions for the duration of the test (~2-3 hours)
* No known contraindications to head movement (e.g., musculoskeletal or neurological conditions that prevent safe head rotation)
* For vestibular dysfunction group: Participants must have a diagnosed vestibular disorder (e.g., vestibular hypofunction, vestibular neuritis, Meniere's disease, labyrinthitis, vestibular migraine, or post-concussive dizziness)
* For control group: Participants must be free from diagnosed vestibular disorders and report no history of balance issues, dizziness, or vertigo

Exclusion Criteria:

* Severe visual impairment that cannot be corrected with glasses or contact lenses
* Cognitive impairment or neurological conditions that could interfere with following instructions (e.g., moderate to severe dementia, uncontrolled seizures, severe traumatic brain injury)
* Severe musculoskeletal or orthopedic conditions affecting the neck or cervical spine that prevent safe head movement (e.g., cervical fusion, severe arthritis, neck instability)
* Acute illness or infection at the time of testing (e.g., flu, COVID-19, severe sinus infection that may impact vestibular function)
* Recent vestibular or neurological surgery (<6 months prior to study participation)
* Severe hearing loss that prevents understanding spoken instructions
* History of stroke or progressive neurological disorders affecting balance or gaze stability (e.g., Parkinson's disease, multiple sclerosis, ALS)
* Use of vestibular suppressants (e.g., meclizine, diazepam, scopolamine) within 24 hours of testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of healthy volunteers employed by or affiliated with the University of Virginia; a convenience sample established patients of the University of Virginia health system who meet study criteria to be subjects in unilateral peripheral vestibular dysfunction (UVD) group
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of mVOR mHealth application system in assessing gaze stability | Immediately after testing (single session, approximately 2-3 hour per participant)
  The mVOR application is expected to be able to distinguish the direction and peak velocity of head rotation as well as the consistency of gaze fixation. The primary outcome measure for this system is the "GST score", which is recorded as the maximum head velocity (in degrees/s) while maintaining visual acuity, a measure of gaze stabilization or dynamic visual. This clinical measure of vestibular function will be compared to a commercially available, in-office system (Bertex, Inc) that utilizes the GST protocol and a head-mounted sensory and is often used in Dizziness and Balance Centers around the world for vestibular rehabilitation.
  Primary variable analysis will include standard descriptive statistics and within-group and between in-group (UVD vs healthy volunteer) pairwise comparisons. ROC and AUC curves will be generated to evaluate the sensitivity and specificity of the mVOR application in distinguishing vestibular dysfunction from healthy controls.

SECONDARY OUTCOMES:
Assessment of static visual acuity | Immediately during (2-3 hours) and following testing
  The mVOR application is expected to be able to distinguish the direction and peak velocity of head rotation as well as the consistency of gaze fixation. In order to do this, per the gaze stabilization test (GST) protocol, the mHealth application must first determine a user's visual acuity with head kept still. This is called the static visual acuity (SVA) and is recorded in logMAR units.
  Primary variable analyses will include standard descriptive statistic and will also be compared to the same outcome measure obtained from a commercially available, in-office GST system.
Assessment of visual perception time | Immediately during (2-3 hours) and following testing
  The mVOR application is expected to be able to distinguish the direction and peak velocity of head rotation as well as the consistency of gaze fixation. In order to do this, per the gaze stabilization test (GST) protocol, the mHealth application .(following determination of the static visual acuity [SVA]), must determine the minimum time at which a user can correctly identify a presented target with head kept still. This outcome measure is called the visual perception time (VPT) and is recorded in milliseconds (msec). Primary variable analyses will include standard descriptive statistic and will also be compared to the same outcome measure obtained from a commercially available, in-office GST system.

OTHER OUTCOMES:
Age | Prior to study enrollment and immediately after testing (single session, approximately 2-3 hour per participant)
  The following user/patient demographic will be obtained either prospectively throughout the clinical trial or retrospectively via the electronic medical record (EMR):
  The subject's age (in years) will be recorded.
  This will be analysed via standard descriptive statistics.
Gender | Prior to study enrollment and immediately after testing (single session, approximately 2-3 hour per participant)
  The following user/patient demographic will be obtained either prospectively throughout the clinical trial or retrospectively via the electronic medical record (EMR):
  The subject's sex (male, female) will be recorded.
  This will be analysed via standard descriptive statistics.
Dizziness Handicap Inventory (DHI) score | Immediately after testing (single session, approximately 2-3 hour per participant)
  The following user/patient demographic will be obtained either prospectively throughout the clinical trial:
  Scores on the validated Dizziness Handicap Inventory (DHI) survey (scale 0-100)
  16-34 Points (mild handicap), 36-52 Points (moderate handicap), and 54+ Points (severe handicap)
  This will be analysed via standard descriptive statistics.
Activities-specific Balance Confidence Scale (ABC Scale) score | Immediately after testing (single session, approximately 2-3 hour per participant)
  The following user/patient demographic will be obtained prospectively throughout the clinical trial:
  Scores on the validated Activities-specific Balance Confidence Scale (ABC Scale) survey (scale 0-100%)
  0% represents no confidence in performing an activity without losing balance and 100% indicates complete confidence
  This will be analysed via standard descriptive statistics
Duration from caloric testing | Prior to study enrollment and immediately after testing (single session, approximately 2-3 hour per participant)
  The following user/patient demographic will be obtained retrospectively via the electronic medical record (EMR):
  Duration from caloric testing (recorded in years), a part of the videonystagmography (VNG) test
  This will be analysed via standard descriptive statistics.
Duration of known vestibular dysfunction | Prior to study enrollment and immediately after testing (single session, approximately 2-3 hour per participant)
  The following patient factor will be retrospectively via the electronic medical record (EMR):
  Duration of known vestibular dysfunction, recorded in years.
  This will be analyzed via standard descriptive statistics.
Side of vestibular dysfunction | Prior to study enrollment and immediately after testing (single session, approximately 2-3 hour per participant)
  The following patient factor will be retrospectively via the electronic medical record (EMR):
  Side of known vestibular dysfunction, recorded as left or right.
  This will be analyzed via standard descriptive statistics.
Duration of vestibular physical therapy | Prior to study enrollment and immediately after testing (single session, approximately 2-3 hour per participant)
  The following patient factor will be retrospectively via the electronic medical record (EMR):
  Duration of vestibular physical therapy, recorded in years
  This will be analyzed via standard descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Thompson-Harvey, MD, Principal Investigator — University of Virginia; Bradley Kesser, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Viginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) will be shared with other researchers upon request. The following data will be made available:
  Demographic Information (age, gender, group allocation - control vs. vestibular dysfunction) Outcome Measures (static visual acuity in logMAR, perception time in ms, maximum head velocity in deg/s) Comparison Data (mVOR mHealth application GST results vs. in-office computerized GST results) Statistical Analysis Outputs (correlation coefficients, ROC curve data, Bland-Altman plots) Data will be shared in compliance with applicable privacy laws and regulations, ensuring that all information remains de-identified and anonymized. Requests for data access will be reviewed by the study investigators and granted for research purposes related to vestibular assessment, gaze stabilization, and telehealth applications.
  Researchers interested in accessing the data may contact the principal investigator.
Time Frame: Start Date: Data and supporting information will be available six months after study completion to allow for initial publication of findings.
  End Date: Data will remain available for at least five years post-publication or as required by funders and institutional policies.
Access Criteria: Who can access the data?
  Qualified researchers, academic institutions, and healthcare professionals conducting research related to vestibular function, gaze stabilization, or telehealth applications.
  What data will be accessible?
  De-identified individual participant data (IPD), including demographic variables, study outcomes, and comparison data between mVOR mHealth application and in-office computerized GST.
  Supporting documents such as the study protocol, statistical analysis plan (SAP), clinical study report (CSR), and analytic code for reproducing study results.
  How to access the data?
  Researchers must submit a formal data request to the principal investigator. Requests will be reviewed on a case-by-case basis to ensure appropriate research use.
  Upon approval, access to datasets and supporting information will be provided through a secure data-sharing repository or via institutional agreements.

REFERENCES:
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Jacobson GP, Newman CW. The development of the Dizziness Handicap Inventory. Arch Otolaryngol Head Neck Surg. 1990 Apr;116(4):424-7. doi: 10.1001/archotol.1990.01870040046011. PMID 2317323
- [Background] Huang K, Sparto PJ, Kiesler S, Siewiorek DP, Smailagic A. iPod-based in-home system for monitoring gaze-stabilization exercise compliance of individuals with vestibular hypofunction. J Neuroeng Rehabil. 2014 Apr 21;11:69. doi: 10.1186/1743-0003-11-69. PMID 24746068
- [Background] Chen PY, Hsieh WL, Wei SH, Kao CL. Interactive wiimote gaze stabilization exercise training system for patients with vestibular hypofunction. J Neuroeng Rehabil. 2012 Oct 9;9:77. doi: 10.1186/1743-0003-9-77. PMID 23043886
- [Background] Goebel JA, Tungsiripat N, Sinks B, Carmody J. Gaze stabilization test: a new clinical test of unilateral vestibular dysfunction. Otol Neurotol. 2007 Jan;28(1):68-73. doi: 10.1097/01.mao.0000244351.42201.a7. PMID 17106431
- [Background] Hall CD, Heusel-Gillig L, Tusa RJ, Herdman SJ. Efficacy of gaze stability exercises in older adults with dizziness. J Neurol Phys Ther. 2010 Jun;34(2):64-9. doi: 10.1097/NPT.0b013e3181dde6d8. PMID 20588090
- [Background] Hall CD, Herdman SJ, Whitney SL, Cass SP, Clendaniel RA, Fife TD, Furman JM, Getchius TS, Goebel JA, Shepard NT, Woodhouse SN. Vestibular Rehabilitation for Peripheral Vestibular Hypofunction: An Evidence-Based Clinical Practice Guideline: FROM THE AMERICAN PHYSICAL THERAPY ASSOCIATION NEUROLOGY SECTION. J Neurol Phys Ther. 2016 Apr;40(2):124-55. doi: 10.1097/NPT.0000000000000120. PMID 26913496
- [Background] Agrawal Y, Carey JP, Della Santina CC, Schubert MC, Minor LB. Disorders of balance and vestibular function in US adults: data from the National Health and Nutrition Examination Survey, 2001-2004. Arch Intern Med. 2009 May 25;169(10):938-44. doi: 10.1001/archinternmed.2009.66. PMID 19468085